CLINICAL TRIAL: NCT06536712
Title: Investigating the Effect of Intraperitoneal Administration of Exosome in Preventing Early Anastomotic Leakage in Rectal Cancer Patients Who Undergo Low Anterior Resection
Brief Title: Effects of Exosome Adminstration in Preventing Early Leakage in Rectal Cancer Patients Undergoing Low Anterior Resection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ahmadi tafti, Assistant professor, Tehran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IR.TUMS.IKHC.REC.1403.114
Record Dates: First submitted 2024-07-20; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells Derived Exosomes (Experimental): 10 patients in this arm will receive Mesenchymal Stem Cells Derived Exosomes at the end of their low anterior resection surgery
  Interventions: Biological: Mesenchymal Stem Cells Derived Exosomes
- Placebo (Placebo Comparator): 10 patients in this arm will receive placebo at the end of their low anterior resection surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal Stem Cells Derived Exosomes — Mesenchymal Stem Cells Derived Exosomes will be administered intraperitoneally to patients at the end of their surgery
  Arms: Mesenchymal Stem Cells Derived Exosomes
Other: Placebo — 10 patients will receive intraperitoneal placebo at the end of their surgery
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of Human Placenta Mesenchymal Stem Cells Derived Exosomes in preventing early anastomosis leak in patients undergoing low anterior resection for rectal cancer. The main question it aims to answer are

Do Mesenchymal Stem Cell-Derived Exosomes prevent early anastomosis leak in patients undergoing low anterior resection for rectal cancer?

If there is a comparison group: Researchers will compare Mesenchymal Stem Cells Derived Exosomes to placebo to see if it can prevent early anastomotic leakage.

Participants will receive intraperitoneal Mesenchymal Stem Cells Derived Exosomes at the end of their surgery.

DETAILED DESCRIPTION:
Anastomotic leakage remains one of the most severe complications following colorectal surgery, leading to increased morbidity, prolonged hospitalization, and reduced quality of life. Despite advances in surgical techniques and perioperative care, the incidence of early anastomotic leaks persists. Practical strategies to reduce this risk are crucial for improving patient outcomes.

Recent studies have highlighted the potential role of mesenchymal stem cell-derived exosomes in enhancing tissue repair and modulating inflammation. These extracellular vesicles, derived from human placenta mesenchymal stem cells (hPMSC), contain bioactive molecules such as proteins, lipids, and RNA that facilitate cellular communication and promote healing processes. Preclinical research suggests that exosomes can support anastomotic healing by reducing local inflammation.

This study aims to evaluate the safety and efficacy of intraperitoneal administration of hPMSC-derived exosomes in preventing early anastomotic leakage in patients undergoing low anterior resection (LAR) for rectal cancer. We hypothesize that the exosome treatment will significantly reduce the incidence of anastomotic leaks compared to placebo, thereby improving postoperative recovery and reducing hospital stay.

ELIGIBILITY:
Inclusion Criteria:

-Patients with Stage II-III rectal cancer who underwent neoadjuvant chemoradiation therapy and are candidates for low anterior resection surgery

Exclusion Criteria:

* Patients who need emergency surgery (presenting with peritonitis or signs of obstruction)
* Patients with apparent malnutrition or patients who have serum albumin levels of less than 3 g/dl
* Patients who receive corticosteroids ( an equivalent dose of prednisolone 5 mg/day or more)
* Patients with chronic pulmonary disease
* Patients who need more than two units of blood transfusion perioperatively

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with early anastomotic leakage | 1 month
  Failed surgical anastomosis after surgery measured with interview and physical examinations in follow-up sessions in clinic

SECONDARY OUTCOMES:
Mean serum and peritoneal Interleukin-6 and Tumor necrosis factor-alpha levels in participants | 1 month
  The level of serum and peritoneal inflammatory markers in postoperative days measured with laboratory tests
Anastomosis integrity in Colonoscopy exam | 1 month
  A colonoscopy will be conducted one month after surgery to assess the integrity of the colorectal anastomosis, detect early signs of local recurrence, identify polyps, and monitor for any postoperative complications such as strictures or inflammatory changes. Baseline colonoscopies will be compared with post-surgical colonoscopy at one month. This outcome will help determine the efficacy of surgical intervention and guide future surveillance strategies in rectal cancer management.
Hospitalization length of stay | 1 month
  The number of days that the patient in hospitalized postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Mohsen Ahmadi Tafti, MD, Study Director — Colorectal Research Center, Imam Khomeini Hospital, Tehran University of Medical Sciences,
Locations (1):
- Division of Colorectal Surgery, Department of Surgery, Tehran University of Medical Sciences, Tehran, Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Platell C, Barwood N, Dorfmann G, Makin G. The incidence of anastomotic leaks in patients undergoing colorectal surgery. Colorectal Dis. 2007 Jan;9(1):71-9. doi: 10.1111/j.1463-1318.2006.01002.x. PMID 17181849
- [Background] Lipska MA, Bissett IP, Parry BR, Merrie AE. Anastomotic leakage after lower gastrointestinal anastomosis: men are at a higher risk. ANZ J Surg. 2006 Jul;76(7):579-85. doi: 10.1111/j.1445-2197.2006.03780.x. PMID 16813622
- [Background] Choi HK, Law WL, Ho JW. Leakage after resection and intraperitoneal anastomosis for colorectal malignancy: analysis of risk factors. Dis Colon Rectum. 2006 Nov;49(11):1719-25. doi: 10.1007/s10350-006-0703-2. PMID 17051321
- [Background] Barnhoorn MC, Wasser MNJM, Roelofs H, Maljaars PWJ, Molendijk I, Bonsing BA, Oosten LEM, Dijkstra G, van der Woude CJ, Roelen DL, Zwaginga JJ, Verspaget HW, Fibbe WE, Hommes DW, Peeters KCMJ, van der Meulen-de Jong AE. Long-term Evaluation of Allogeneic Bone Marrow-derived Mesenchymal Stromal Cell Therapy for Crohn's Disease Perianal Fistulas. J Crohns Colitis. 2020 Jan 1;14(1):64-70. doi: 10.1093/ecco-jcc/jjz116. PMID 31197361
- [Background] Tashak Golroudbari H, Banikarimi SP, Ayati A, Hadizadeh A, Khorasani Zavareh Z, Hajikhani K, Heirani-Tabasi A, Ahmadi Tafti M, Davoodi S, Ahmadi Tafti H. Advanced micro-/nanotechnologies for exosome encapsulation and targeting in regenerative medicine. Clin Exp Med. 2023 Oct;23(6):1845-1866. doi: 10.1007/s10238-023-00993-7. Epub 2023 Jan 27. PMID 36705868